CLINICAL TRIAL: NCT04336501
Title: Efficacy Study About Donor Derived CD19-target T Cell to Treat B-ALL Post Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy and Safety Evaluation of IM19 CAR-T Cell Therapy for MRD+ After Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART20190423
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CAR-T group (Experimental): Subject will be treated with IM19 car-t cells
  Interventions: Biological: IM19 CAR-T

INTERVENTIONS:
Biological: IM19 CAR-T — All patients will be treated with fludarabine and cyclophosphamide for 3 days,then,CAR-T cells expressing CD19 CAR will be infused 24-96 hours later

SUMMARY:
Efficacy study about donor derived CD19-target T cell to treat B-ALL post hematopoietic stem cell transplantation

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-hsct) for the treatment of refractory recurrent acute b-lymphoblastic leukemia (b-all), the overall survival rate of 3 years after transplantation was about 10%. The overall survival rate at 3 years was about 70 percent. In the early stage, the investigators established the monitoring method of leukemia micro-residual disease, effectively screened out the high-risk group of recurrence, combined with the new relapse treatment method, successfully implemented the stratification and even personalized dry prediction of leukemia recurrence for the first time in the world, and reduced the recurrence rate of the high-risk group by 30%. However, the therapeutic targeting is not strong, and up to 30% of patients will develop graft versus host disease, which seriously affects the survival of patients. The use of CAR repair T cells (CAR T) to target CD19 in the treatment of refractory recurrent b-all was effective, and the use of CAR T in the treatment of recurrent b-all after transplantation did not increase the risk of GVHD. This clinical study mainly discussed the safety and efficacy of donor targeted cd19-t cells after allo-hsct in the treatment of acute b-lymphocytic leukemia with minimal residual disease. It is expected that the recurrence rate will be reduced while the incidence of acute GVHD after transplantation will not be increase

ELIGIBILITY:
Inclusion Criteria:

* To be aged 3 to 65 years
* It was consistent with the diagnosis of CD19+ B-All with MRD+ in allo- hsct transplantation
* The immunotyping was determined to be CD19+ B-All
* The T lymphocytes in the subjects were 100% donor T lymphocytes
* No chemotherapy or antibody treatment was received 2 weeks before cell therapy
* Left ventricular ejection fraction (LVEF) ≥50% and centerless inclusion were diagnosed by echocardiography
* The subjects had no pulmonary active infection
* Blood oxygen saturation at the fingertips ≥ 92%
* Estimated survival of >3 months
* ECOG physical condition level 0~1

Exclusion Criteria:

* Unwilling to accept IM19 CAR-T cell therapy, do not agree to signInformed consent of subject
* Subjects are allergic to the components of cellular products
* Total serum bilirubin ≥ 2.0mg/dl、Serum albumin < 35g/L、ALT and AST were more than 3 times of the upper limit of the normal range. Blood creatinine ≥ 2.0mg/dl;Platelet < 20 x 109 / L
* Subjects had activity level II-IV aGVHD, or activityModerate to severe cGVHD
* The subjects had a severe failure to control the infection
* Subject with known central nervous system leukemia (CNS2 or CNS3)
* Subjects were treated with CAR T cells or DLT after transplantation
* The subjects developed bone marrow failure syndrome after allo-hsct transplantation
* The subjects had previously received other gene treatments
* The subjects had a history of alcohol, drug use or mental illness
* Subjects were enrolled in any other clinical investigator within 1 month prior to screening
* Female subjects: 1) were pregnant/lactating, or 2) had a pregnancy plan during the study period,Or 3) fertile and unable to use effective contraception
* The researchers believe there are other conditions that may not be appropriate for the study

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR at 6 month | 6 months
  Objective response at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: xiang yu zhao, MD, Principal Investigator — Peking University people's hospita
Locations (1):
- Peking University people's hospita, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No